CLINICAL TRIAL: NCT04261465
Title: The NUVOLA TRIAL: Neoadjuvant Chemotherapy in Unresectable oVarian Cancer With OLAparib and Weekly Carboplatin Plus Paclitaxel: A Phase II Open-label Multicentre Study
Brief Title: NUVOLA TRIAL Open-label Multicentre Study
Acronym: NUVOLA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2345
Record Dates: First submitted 2020-01-31; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-11

CONDITIONS: High Grade Serous Ovarian Cancer
MeSH Terms: interventions — olaparib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel Carboplatin Olaparib (Experimental): Subjects will receive weekly therapy with paclitaxel 60 mg/m2 IV and carboplatin AUC 2 IV for 3 weeks out of 4, and olaparib tablets at the dose of 150 mg bid administered orally for 3 consecutive days (D1-D3), every week for each cycle.
  After 3 cycles patients will be evaluated for interval debulking surgery. After surgery they will receive consolidation treatment with paclitaxel and carboplatin according to Investigator's choice
  Interventions: Drug: Olaparib; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Olaparib — PARP INHIBITOR
  Other Names: Lynparza
Drug: Paclitaxel — Chemotherapy
Drug: Carboplatin — Chemotherapy

SUMMARY:
Around 15-25% of ovarian cancer (OC) patients carry germ-line mutation in BRCA1 or BRCA2 genes. Recent evidences showed that OC women with germline BRCA1/2 mutations (gBRCAmut) have an improved survival and higher platinum-sensitivity compared to BRCA1/2 naive (BRCAwt).

Interestingly, disease appearance in BRCAmut women is more diffuse than in BRCAwt cases, with significantly higher peritoneal tumour load.

Nonetheless, BRCAmut women additionally show a higher benefit of platinum-based neoadjuvant chemotherapy (NACT) plus interval debulking surgery compared with BRCAwt women in terms of clinical and pathological responses, suggesting that BRCA mutational status might be used as a molecular tool to personalize treatment in high-grade serous ovarian cancer (HGSOC) patients.

OLAPARIB in BRCA mutation carriers Olaparib is a potent oral poly (ADP-ribose) polymerase (PARP) inhibitor that causes synthetic lethality in BRCA1/2-deficient tumour cells. In patients with platinum-sensitive relapsed serous ovarian cancer, olaparib maintenance treatment significantly improved the duration of progression-free survival compared with placebo (hazard ratio [HR] 0.35 [95% CI (confidence interval) 0.25-0.49]; p<0.0001), with the greatest clinical benefit in patients with BRCA mutations (HR 0.18 [95% CI 0.10-0.31]; p<0.0001).

Preclinical data suggest that olaparib might also potentiate the efficacy of DNA-damaging chemotherapies, including platinum-containing drugs such as carboplatin.

In a recent phase Ib/II study, olaparib plus weekly carboplatin and paclitaxel in relapsed ovarian cancer patients was shown to be safe, well tolerated and effective, especially in germline BRCA mutated (gBRCAmut) patients.

Possibly, the addition of a PARP inhibitor (olaparib) to NACT in HGSOC patient with germline or somatic BRCA1/2 mutation is able to increase the pathological complete response rate to conventional chemotherapy. Combination of intermittent olaparib with weekly carboplatin and paclitaxel might achieve a higher pathological response rate, with an acceptable toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed advanced high grade serous or endometrioid ovarian, fallopian tube, or primary peritoneal cancer;
2. Female, aged at least 18 years;
3. Documented mutation in BRCA1 or BRCA2 germline and/or somatic that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function);
4. FIGO stages III-IV primary ovarian, primary peritoneal, or fallopian tube cancers not suitable of primary cytoreductive surgery (Criteria for Neoadjuvant Chemotherapy despite to Primary Surgery: clinical conditions; Fagotti's score > 10, small bowel carcinosis, mesenteric retraction);
5. Measurable disease according to RECIST criteria 1.1;
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
7. Left Ventricular Ejection Fraction (LVEF) ≥ institutional lower limit of normal;
8. Patients must have a life expectancy of >16 weeks;
9. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   1. Haemoglobin ≥ 10.0 g/dL and no blood transfusions in the 28 days prior to entry/randomisation (choose whichever is most applicable to the study)
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   3. No features suggestive of MDS/AML on peripheral blood smear
   4. White blood cells (WBC) > 3x109/L
   5. Platelets count ≥ 100 x 109/L
   6. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   7. AST (Aspartate Aminotransferase)/ALT (Alanine aminotransferase) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   8. Creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min using the Cockcroft-Gault equation.

   Estimated creatinine clearance =[ (140-age [years]) x weight (kg) (x F)] /[serum creatinine (mg/dL) x 72]; where F=0.85 for females
10. No other invasive malignancy within the past 3 years except non-melanoma skin cancer or in situ cervical cancer (patients with previous cancers may be enrolled providing that no recurrences have be reported in the last 3 years);
11. Written Informed Consent;
12. Postmenopausal status defined as:

    Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50 Radiation-induced oophorectomy with last menses >1 year ago Chemotherapy-induced menopause with >1 year interval since last menses Surgical sterilisation (bilateral oophorectomy or hysterectomy) or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test prior to Myriad BRCA test during screening part 1, within 28 days of study treatment and confirmed prior to treatment on day 1;
13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations;
14. For inclusion in the optional exploratory genetic and the optional biomarker research, patients must provide informed consent for genetic and for biomarker research

Exclusion Criteria:

1. History of another neoplastic disease (except basal cell carcinoma or cervical carcinoma in situ adequately treated) unless in remission for 5 years or longer
2. Other serious illnesses, such as:

   Congestive heart failure or angina pectoris; myocardial infarction within 3 months before enrolment; uncontrolled arterial hypertension or arrhythmias Psychiatric disorder that prevents compliance with protocol Uncontrolled seizures Active viral hepatitis; or chronic liver disease Active infection Any other unstable medical conditions
3. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
4. Non defective BRCA status or BRCA 1 and/or BRCA2 mutations that are considered to be non detrimental (e.g."Variants of uncertain clinical significance" or "Variant of unknown significance"or "Variant, favor polymorphism" or "benign polymorphism" etc)
5. Patients with early stage disease (FIGO Stage I, IIA, IIB or IIC)
6. Patients who have previously received chemotherapy or radiotherapy for any abdominal or pelvic tumour, including treatment for prior diagnosis at an earlier stage for their ovarian, fallopian tube or primary peritoneal cancer. (Patients who have received prior adjuvant chemotherapy for localised breast cancer may be eligible, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease).
7. Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, unless all of the following conditions are met: Stage not greater than I-A; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO Grade 3 lesions.
8. Participation in another clinical study with an investigational product
9. Any previous treatment with PARP inhibitor, including olaparib.
10. Resting ECG with QTc (corrected QT interval) > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
11. Concomitant use of known potent CYP3A4 (Cytochrome P450 3A4)inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir. The required washout period prior to starting olaparib is 2 weeks.
12. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2 caused by previous cancer therapy, excluding alopecia.
13. Patients with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML.
14. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
15. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
16. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication, including gastrectomy.
17. Breast feeding women.
18. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
19. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
20. Patients with a known hypersensitivity to Paclitaxel or Carboplatin, or any of the excipients of these agents
21. Previous allogeneic bone marrow transplant, or double umbilical cord blood transplantation
22. Previous enrolment in the present study
23. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
24. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents.
25. Whole blood transfusions in the last 120 days prior to entry to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 28 months
  Pathological complete response after 3 cycles of NACT including Olaparib and weekly Carboplatin-Paclitaxel in BRCAmut advanced HGSOC women.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Prof, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Derived] Marchetti C, Tudisco R, Salutari V, Pietragalla A, Scambia G, Fagotti A. Neoadjuvant chemoteraphy in unresectable ovarian cancer with olaparib and weekly carboplatin plus paclitaxel: a phase II, open label multicenter study (NUVOLA trial). Int J Gynecol Cancer. 2021 Aug;31(8):1175-1178. doi: 10.1136/ijgc-2021-002727. Epub 2021 Jun 15. PMID 34131041